CLINICAL TRIAL: NCT02335814
Title: Phase 1/1b, First-in-Human, Dose-Escalation and Expansion Study of FLX925 Administered Orally to Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: First-in-Human Study of FLX925 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose escalation completed; Sponsor decision
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLX925-01
Record Dates: First submitted 2015-01-05; First posted 2015-01-12 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLX925 (Experimental)
  Interventions: Drug: FLX925

INTERVENTIONS:
Drug: FLX925

SUMMARY:
This first-in-human (FIH) clinical trial is a Phase 1/1b, open-label, sequential-group, dose-escalation and cohort expansion study evaluating the safety, PK, PD, and antitumor activity of FLX925 in subjects with relapsed or refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥ 18 yrs;
2. Subjects with histologically confirmed relapsed or treatment refractory AML with the exception of subjects who are in first relapse following a remission >12 months in duration and are eligible for standard therapies (e.g., chemotherapy or stem cell transplantation).
3. Assessment of FLT3 mutation status;
4. Part 2 (Expansion) only: Subject must be able to be stratified into 1 of 3 cohorts:

   * Cohort A: Subjects with a FLT3 mutation (e.g. ITD or D835) with prior FLT3 inhibitor treatment
   * Cohort B: Subjects with a FLT3 mutation (e.g. ITD or D835) without prior FLT3 inhibitor treatment
   * Cohort C: Subjects without a FLT3 mutation at the time of enrollment
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
6. Considered by the investigator to be an appropriate candidate for a Phase 1 clinical study;
7. The interval from prior treatment to time of initiation of FLX925 administration will be ≥ 2 weeks for cytotoxic agents and ≥ 5 half-lives for investigational/non-cytotoxic agents. For patients with rapidly proliferative disease, use of hydroxyurea is allowed if started prior to initiation of study therapy;
8. Clinically significant toxic effects of any prior antitumor therapy (except hydroxyurea) resolved to Grade ≤ 1 before the start of study therapy (bone marrow parameters [Grade 1 to 4 permitted]);
9. Serum AST and ALT ≤ 3 x ULN;
10. Serum bilirubin ≤ 2 x ULN unless due to Gilbert's syndrome or hemolysis or considered to be related to leukemia;
11. Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance (CrCl) of ≥ 60 mL/hour by the Cockroft-Gault equation;
12. Normal coagulation profile as evidenced by PT and aPTT ≤ 1.5 x ULN;
13. For women of childbearing potential, negative serum pregnancy test;
14. Women of childbearing potential and sexually mature males must agree to use a medically accepted method of contraception throughout the study and for 30 days following the last dose;
15. Ability to swallow tablets without difficulty;
16. Willingness to comply with scheduled visits, drug administration plan, protocol-specified bone marrow biopsies;
17. Written informed consent must be provided.

Exclusion Criteria:

1. Subjects with AML in their first relapse following a remission >12 months in duration who are eligible for standard therapies (e.g. chemotherapy or stem cell transplantation);
2. Absolute leukemic blast count in peripheral blood >50,000/ microliter;
3. Active, symptomatic central nervous system (CNS) leukemia;
4. History of another malignancy except for the following: adequately treated local non-melanoma skin cancer; in situ cervical carcinoma; adequately treated, papillary, non-invasive bladder cancer; asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥ 1 year prior to start of study therapy; other adequately treated Stage 1 or 2 cancers currently in complete remission, or any other cancer that has been in complete remission for ≥ 2 years.
5. Clinically significant cardiovascular disease;
6. Significant screening electrocardiogram (ECG) abnormalities;
7. Significant risk for bleeding due to active peptic ulcer disease or bleeding diathesis or requirement for systemic anticoagulation or history of significant gastrointestinal, urological, intracranial or other significant bleeding within 1 year from the start of treatment;
8. Significant active gastrointestinal disease that might impair absorption of study therapy;
9. Evidence of an ongoing, uncontrolled systemic infection or an uncontrolled local infection requiring therapy at the time of start of study therapy
10. Known or suspected human immunodeficiency virus (HIV) infection or patients who are HIV seropositive;
11. Patients known to be positive for hepatitis B or to have active hepatitis C infection;
12. Any evidence of ongoing graft-versus-host disease (GVHD) in subjects with prior progenitor cell transplantation;
13. Pregnancy or breastfeeding;
14. Major surgery within 4 weeks before the start of study therapy;
15. Ongoing immunosuppressive therapy within 14 days prior to the start of study therapy;
16. Subjects currently receiving treatment with any medications that have the following potential properties and who cannot be either discontinued or switched to a different medication:

    * the potential to prolong the QT interval, or
    * strong CYP3A4 inhibitors, or
    * CYP3A4 or CYP2C19 or P glycoprotein (P-gp) or breast cancer resistance protein (BCRP) substrates having a narrow therapeutic index;
17. Concurrent participation in another therapeutic clinical trial;
18. Any condition deemed by the investigator to be likely to interfere with a subject's ability to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 30 Months
Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of FLX925 | 12 Months
Assess the antitumor activity of FLX925 when administered at the RP2D dose | 30 Months

SECONDARY OUTCOMES:
Evaluate the PK profile of FLX925 (maximum concentration (Cmax), time of the maximum measured concentration (Tmax), area under the concentration-time curve (AUC), and terminal elimination half-life (t1/2) | 30 Months
  PK parameters include: maximum concentration (Cmax), time of the maximum measured concentration (Tmax), area under the concentration-time curve (AUC), and terminal elimination half-life (t1/2)
Assess the effects of FLX925 on pharmacodynamic (PD) markers (changes in FLT3-ITD and FLT3-D835 allelic burden) | 30 Months
  PD endpoints include: changes in FLT3-ITD and FLT3-D835 allelic burden, status and changes in the cyclin/CDK/Rb pathway, and changes in immune parameters
Characterize tumor control according to clinical disease response assessments per Cheson criteria in subjects receiving FLX925 | 30 Months
Explore the relationships of PK and PD parameters to clinical drug activity as defined by clinical disease response assessments per Cheson criteria | 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (12):
- United States (12):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington